CLINICAL TRIAL: NCT02877407
Title: A Randomized Controlled Study of Laparoscopic/Robotic-assisted Hysteropexy Versus Vaginal Hysterectomy for the Treatment of Uterovaginal Prolapse
Brief Title: Laparoscopic/Robotic-assisted Hysteropexy Versus Vaginal Hysterectomy for the Treatment of Uterovaginal Prolapse
Acronym: PROLAPSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Dong Hoon Suh, associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-1605/345-002
Record Dates: First submitted 2016-08-16; First posted 2016-08-24 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Uterovaginal Prolapse; Hysteropexy

ARMS (2):
- laparoscopic/robotic-assisted hysteropexy (Other): patient who undergo laparoscopic/robotic-assisted hysteropexy
  Interventions: Procedure: patient who undergo laparoscopic/robotic-assisted hysteropexy
- vaginal hysterectomy (Other): patient who undergo vaginal hysterectomy
  Interventions: Procedure: patient who undergo vaginal hysterectomy

INTERVENTIONS:
Procedure: patient who undergo laparoscopic/robotic-assisted hysteropexy
  Arms: laparoscopic/robotic-assisted hysteropexy
Procedure: patient who undergo vaginal hysterectomy
  Arms: vaginal hysterectomy

SUMMARY:
* objective: aimed to compare laparoscopic/robot-assisted hysteropexy with vaginal hysterectomy for uterine prolapse
* prospective randomized clinical trial
* patient

  1. 60yrs or more women and
  2. POP-Q stage II with symptom or POP-Q III, IV regardless of symptom
* number of patient: 146
* randomize: laparoscopic/robot-assisted hysteropexy vs. hysterectomy
* follow up: postoperative 1 year
* primary endpoint: recurrence rate

  1. recurrence of uterovaginal prolapse POP-Q stage II-IV
  2. recurrence of associated symptom
* secondary endpoint

  1. postoperative 1 year QOL, degree of satisfaction evaluation
  2. operative time, estimated blood loss
  3. hospitalization period, postoperative pain, return to normal activity

ELIGIBILITY:
Inclusion Criteria:

* POP-Q stage II with symptom or POP-Q III, IV regardless of symptom

Exclusion Criteria:

* abnormal uterine bleeding
* significantly enlarged fibroid uterus
* postmenopausal uterine bleeding
* endometrial pathology
* on tamexifen
* concomitant medical problems precluding general anesthesia or surgery
* damaged agreement ability

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
recurrence rate (%) | postoperative 1 year
  recurrence rate(%) of uterovaginal prolapse POP-Q stage II-IV in postoperative 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dong Hun Suh, associate professor, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National Univesity Bundang Hospital, Seongnam-si, Kyeonggi-do, South Korea